CLINICAL TRIAL: NCT01753648
Title: Non-invasive Measurement of Retinal Blood Flow Based on Vessel Analysis and Fourier Domain Optical Coherence Tomography in Patients With Hypertensive Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-220612
Record Dates: First submitted 2012-12-07; First posted 2012-12-20 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Hypertensive Retinopathy
Keywords: retinal blood flow; retinal blood velocity; retinal oxygen saturation; retinal vessel diameter; ocular perfusion pressure
MeSH Terms: conditions — Hypertensive Retinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertensive retinopathy (Experimental): 30 patients with hypertensive retinopathy stage 2 or 3
  Interventions: Device: Dynamic Vessel Analyzer; Other: FDOCT; Other: Ocular perfusion pressure
- healthy controls (Experimental): 30 healthy age- and sex-matched controls
  Interventions: Device: Dynamic Vessel Analyzer; Other: FDOCT; Other: Ocular perfusion pressure

INTERVENTIONS:
Device: Dynamic Vessel Analyzer — Retinal vessel diameter, total retinal blood flow (together with FD-OCT), retinal oxygen saturation
Other: FDOCT — total retinal blood flow (together with DVA), retinal blood velocities
  Other Names: Fourier Domain Color Doppler Optical Coherence Tomography
Other: Ocular perfusion pressure — Measurement of intraocular pressure and mean arterial blood pressure for determination of ocular perfusion pressure

SUMMARY:
Recently, a new and sophisticated method for assessment of retinal blood flow and retinal blood flow velocity profiles has become available. This technique is based on the combination of measurement of retinal vessel calibers with bidirectional Fourier domain optical coherence tomography (FDOCT). The valid measurement of retinal blood flow is of significant importance, because it is known that major ophthalmic diseases, such as hypertensive retinopathy, are associated with alterations in blood flow.

Hypertensive retinopathy is the most common manifestation of arterial hypertension in the eye. Elevated systemic blood pressure leads to generalized arteriolar narrowing caused by vasospasms and increased vascular tone. Further in the disease process, focal arteriolar narrowing, retinal haemorrhages, hard exudates and cotton wool spots can occur. Previous studies have shown that blood flow in the extraocular vessels and in the choroid is compromised in patients with arterial hypertension. However, data on the impact of arterial hypertension on retinal blood flow and retinal blood flow velocities are lacking.

The present study sets out to compare total retinal blood flow and retinal velocity profiles in patients with hypertensive retinopathy and healthy age- and sex-matched controls. Ocular perfusion pressure will be calculated based on measurements of blood pressure and intraocular pressure to allow for calculation of vascular resistance. In addition, velocity profiles at arterio-venous crossings will be measured. It is hypothesized that these velocity profiles are considerably modified in patients with stage 2 and 3 hypertensive retinopathy compared to healthy controls because of pronounced arterio-venous compression.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects

* Men and women aged over 18 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Systolic Blood Pressure ≤ 120 mmHg and Diastolic Blood Pressure ≤ 80 mmHg
* Normal ophthalmic findings, ametropia < 6 Dpt.

Inclusion criteria for patients with hypertensive retinopathy

* Men and women aged over 18 years
* Hypertensive retinopathy stage 2 or 3
* Normal ophthalmic findings except hypertensive retinopathy stage 2 and 3, ametropia < 6 Dpt.

Exclusion Criteria:

Any of the following will exclude a healthy subject from the study:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Presence or history of arterial hypertension
* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study (except oral contraceptive)
* Blood donation during the previous three weeks
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Ametropia >= 6 Dpt
* Pregnancy, planned pregnancy or lactating

Any of the following will exclude a patient with hypertensive retinopathy from the study:

* Participation in a clinical trial in the 3 weeks preceding the screening visit
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Blood donation during the previous three weeks
* Hypertensive retinopathy stage 4
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Ametropia >= 6 Dpt
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Total retinal blood flow | 1 day

SECONDARY OUTCOMES:
Retinal vessel diameter | 1 day
Retinal blood velocities | 1 day
Ocular perfusion pressure | 1 day
Retinal (arterial and venous) oxygen saturation | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria